CLINICAL TRIAL: NCT07247942
Title: A Phase I, Open-label Study of the Metabolism and Excretion of [14C]-Zidebactam (WCK 5107) Following a Single Intravenous Infusion in Healthy Male Subjects.
Brief Title: Study of the Metabolism and Excretion of Zidebactam (WCK 5107) Following a Single Intravenous Infusion.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wockhardt (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: W-5107-103
Record Dates: First submitted 2025-09-23; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Healthy Subjects (HS)
Keywords: zidebactam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- zidebactam administered as a 1g (approximately 200 μCi) IV infusion over 1 hour (Experimental)
  Interventions: Drug: zidebactam administered as a 1g (approximately 200 μCi) IV infusion over 1 hour

INTERVENTIONS:
Drug: zidebactam administered as a 1g (approximately 200 μCi) IV infusion over 1 hour — zidebactam administered as a 1g (approximately 200 μCi) IV infusion over 1 hour following at least an 8-hour fast from food (not including water).

SUMMARY:
A Phase 1, Open-label Study of the Metabolism and Excretion of Zidebactam (WCK 5107) Following a Single Intravenous Infusion in Healthy Male Subjects

DETAILED DESCRIPTION:
The primary objectives of the study are:

* To determine mass balance and routes of elimination of [zidebactam following administration of a single 1g (approximately 200 μCi) radiolabeled intravenous (IV) infusion of zidebactam in healthy male subjects
* To assess the pharmacokinetics (PK) of a single IV infusion of zidebactam
* To determine the whole blood and plasma concentrations of total radioactivity following a single IV infusion of -zidebactam
* To determine the urinary and fecal recovery of the total administered radioactive dose

The secondary objectives of the study are:

* To characterize and identify metabolites of zidebactam in plasma, urine, and feces, as applicable
* To determine plasma and urine concentrations of non-radiolabeled zidebactam
* To assess the safety and tolerability of zidebactam

ELIGIBILITY:
Inclusion Criteria:

* 1. Body mass index between 18.5 and 29.9 kg/m2, inclusive at Screening and Check-in (Day -1).

  2. In good health, determined by no clinically significant findings from medical history, physical examination (at Check-in [Day -1]), 12-lead ECG, vital signs measurements, and clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia [eg, Gilbert's syndrome] is not acceptable) at Screening or Check-in as assessed by the Investigator (or designee).

  3. Blood pressure between 90 and 140 mmHg systolic, inclusive, and not higher than 90 mmHg diastolic, unless deemed not clinically significant by the Investigator (or designee).

  4. History of a minimum of 1 bowel movement per day.

Exclusion Criteria:

* 1. Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder.

  2. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance.

  3. History of alcoholism or drug/chemical abuse within 1 year prior to Check-in (Day -1).

  4. Alcohol consumption of >28 units per week for males. One unit of alcohol equals 12 oz. (360 mL) of beer, 1½ oz. (45 mL) of liquor, or 5 oz. (150 mL) of wine.

  5. Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's Wort, within 14 days prior to Check-in.

  6. Subjects with exposure to significant diagnostic or therapeutic radiation (eg, serial X-ray, computed tomography scan, barium meal) or current employment in a job requiring radiation exposure monitoring within 12 months prior to Check-in.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 8 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2018-01-20 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Amount Excreted in Urine (Aeu) | 7 days
  The primary PK outcome endpoints of zidebactam and total radioactivity derived from urine collections is the amount excreted in urine (Aeu).
Cumulative Aeu in urine (Cum Aeu) | 7 days
  The primary PK outcome endpoints of zidebactam and total radioactivity derived from urine collections is the cumulative Aeu (Cum Aeu).
Percentage excreted in urine (feu): | 7 days
  The primary PK outcome endpoints of zidebactam and total radioactivity derived from urine collections is the percentage excreted in urine (feu).
Cumulative feu in urine(Cum feu): | 7 days
  The primary PK outcome endpoints of zidebactam and total radioactivity derived from urine collections is the cumulative feu (Cum feu).
Renal clearance (zidebactam only; CLR): | 7 days
  The primary PK outcome endpoints of zidebactam and total radioactivity derived from urine collections is the renal clearance (zidebactam only; CLR).
Amount excreted in feces (Aef): | 7 days
  The primary PK outcome endpoints of total radioactivity derived from fecal collections were the amount excreted in feces (Aef).
Cumulative Aef in feces (Cum Aef): | 7 days
  The primary PK outcome endpoints of total radioactivity derived from fecal collections were the cumulative Aef (Cum Aef).
Percentage excreted in feces (fef): | 7 days
  The primary PK outcome endpoints of total radioactivity derived from fecal collections were the percentage excreted in feces (fef).
Cumulative fef in feces (Cum fef): | 7 days
  The primary PK outcome endpoints of total radioactivity derived from fecal collections were the cumulative fef (Cum fef).

SECONDARY OUTCOMES:
Metabolic Profile of [14C]-zidebactam | 7 days
  The secondary metabolite endpoints is the metabolic profile of [14C]-zidebactam
Identification of [14C]-zidebactam metabolites | 7 days
  The identification of [14C]-zidebactam metabolites is a secondary metabolite endpoint.
Incidence and severity of AEs | 7 Days
  The incidence and severity of adverse events (AEs) is a secondary safety outcome measure.
Incidence of laboratory abnormalities, based on hematology, clinical chemistry, coagulation, and urinalysis test results | 7 days
  The incidence of laboratory abnormalities, based on hematology, clinical chemistry, coagulation, and urinalysis test results, is a secondary safety outcome measure.
12-lead electrocardiogram (ECG) parameters | 7 days
  The assessment of 12-lead electrocardiogram ECG QT Interval parameters is included as a secondary safety outcome measure.
Vital Signs -Supine Blood Pressure | 7 days
  Supine Blood Pressure is a secondary outcome measure
Physical Examinations | 7 days
  Physical examinations is a secondary safety outcome measure. To assess the outcome measure a questionnaire includes below mentioned measurements.
  General Appearance Skin Lymph Nodes HEENT Neck Thorax/Lungs Cardiovascular Abdomen Musculoskeletal Neurological
Vital Signs- supine pulse rate | 7 days
  supine pulse rate is a secondary outcome measure
Vital Signs- respiratory rate | 7 Days
  respiratory rate is a secondary outcome measure
Vital signs- oral body temperature | 7 days
  oral body temperature is a secondary outcome measure

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Clinical Research Unit Inc. 3402 Kinsman Boulevard Madison, Wisconsin 53704 USA, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2017-11-13): https://cdn.clinicaltrials.gov/large-docs/42/NCT07247942/Prot_000.pdf
  • Informed Consent Form (2017-11-20): https://cdn.clinicaltrials.gov/large-docs/42/NCT07247942/ICF_001.pdf